CLINICAL TRIAL: NCT07013565
Title: NYMC623: A Comprehensive Risk-adapted Chemommunotherapy Protocol of Emerging Immunotherapies for Relapsed/Refractory Alk+ Anaplastic Large Cell Lymphoma (ACCELERATE)
Brief Title: Chemoimmunotherapy for ALK+ Relapsed/Refractory ALCL
Acronym: ACCELERATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: University of Alabama at Birmingham (Other); Helen DeVos Children's Hospital (Other); Nationwide Children's Hospital (Other); Memorial Sloan Kettering Cancer Center (Other); University of Utah (Other); Ohio State University (Other); University of North Carolina (Other); Children's Hospital of Philadelphia (Other); Medical College of Wisconsin (Other); Children's Hospital of Orange County (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 623
Record Dates: First submitted 2025-05-06; First posted 2025-06-10 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Positive
Keywords: ALCL; Relapsed ALCL
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic | interventions — Vinblastine; Brentuximab Vedotin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low-risk ALK+ ALCL (Experimental): Low risk patients include any patient with FIRST RELAPSE > ONE YEAR from initial diagnosis of de novo ALK+ ALCL,Common histology, CD3 negative, Minimum disseminated disease (MDD) negative at de novo diagnosis (if MDD known), AND No prior exposure to vinblastine (VBL).
  Interventions: Drug: Vinblastine (Velban)
- High Risk ALK+ ALCL (BV Naive) (Experimental): * Any patient with RELAPSED OR PROGRESSIVE DISEASE ONE YEAR from initial diagnosis of de novo ALK+ ALCL,
  * Small cell/histiocytic histology,
  * CD3 positive (homogeneous staining of CD3 positive T-cells)
  * Second or later relapse,
  * Induction failure during initial treatment for de novo ALK+ ALCL, OR
  * Minimal disseminated disease (MDD) positive at de novo diagnosis (if MDD known)
  Interventions: Drug: Vinblastine (Velban); Drug: Brentuximab vedotin (Adcetris); Drug: Nivolumab (Opdivo)
- High Risk ALK+ ALCL (with prior BV) (Experimental): * Any patient with RELAPSED OR PROGRESSIVE DISEASE ONE YEAR from initial diagnosis of de novo ALK+ ALCL,
  * Small cell/histiocytic histology,
  * CD3 positive (homogeneous staining of CD3 positive T-cells)
  * Second or later relapse,
  * Induction failure during initial treatment for de novo ALK+ ALCL, OR
  * Minimal disseminated disease (MDD) positive at de novo diagnosis (if MDD known)
  Interventions: Drug: Vinblastine (Velban); Drug: Brentuximab vedotin (Adcetris); Drug: Nivolumab (Opdivo)

INTERVENTIONS:
Drug: Vinblastine (Velban) — Low risk cohort patients will receive 2 cycles of Induction therapy with single-drug vinBLAStine (VBL), then undergo disease assessment. If complete remission (CR) and MRD -, LR patients will continue single-drug VBL for a total of 24 months (if absent disease progression or unacceptable toxicity).
Drug: Brentuximab vedotin (Adcetris) — HR cohort patients with no previous exposure to BV will receive 2 cycles of Induction therapy with BV and NIVO [BV + NIVO] one every 21 days, then undergo disease assessment. Patients in CR will proceed with consolidation with RTC allogeneic SCT (SCT)*. If patient has any response other than CR and MRD-, they will receive 2 cycles of BV, VBL, and NIVO [BV + VBL + NIVO] once every 21 days
  Other Names: Nivolumab
  Arms: High Risk ALK+ ALCL (BV Naive); High Risk ALK+ ALCL (with prior BV)
Drug: Nivolumab (Opdivo) — High risk cohort patients with previous exposure to Brentuximab vedotin (BV) will receive 2 cycles of Induction therapy with VBL and NIVO [VBL + NIVO] on day 1 and 15, then undergo disease assessment. If response is not CR, or patient has PR/SD/PD, patient will receive [BV+VBL+NIVO] and subsequent therapy as defined for the HR2 cohort.
  Other Names: brentuximab vedodin; Vinblastine
  Arms: High Risk ALK+ ALCL (BV Naive); High Risk ALK+ ALCL (with prior BV)

SUMMARY:
Children, adolescents, and young adults (CAYA) with relapsed/refractory (R/R) high-risk ALK+ Anaplastic Large Cell Lymphoma (ALCL) have a low incidence of overall survival. This clinical trial will investigate if a new FDA approved medication called Nivolumab (NIVO) (which is a checkpoint blockade immunotherapy) combined with chemotherapy based on the patients risk status to get the patient into the best response possible. Then patients will receive lower doses of chemoimmunotherapy and allogeneic stem cell transplantation (stem cells from another person). The investigators this this new treatment will improve survival rates in this high-risk population of patients.

DETAILED DESCRIPTION:
Brief Background: A multitude of chemotherapeutic regimens have been evaluated for the treatment of de novo ALK+ ALCL. Unfortunately, no chemotherapeutic regimen has improved the 20-30% treatment failure rate. Given the ubiquitous cell surface expression of CD30 on ALK+ ALCL, the anti-CD30 antibody drug conjugate (ADC) brentuximab vedotin (BV) is a rational therapeutic agent for ALK+ ALCL. 16. In the most recent Children's Oncology Group (COG) trial for de novo ALK+ ALCL (ANHL12P1), BV was combined with ALCL99 chemotherapy and demonstrated the best reported outcomes with a 2-year event free survival and overall survival of 79% and 97% respectively. Immune checkpoint inhibition with antibodies that block the inhibitory immune receptors CTLA-4, PD-1, and PD-L1 have improved the outcomes for many patients with cancer by dramatically enhancing the anti-tumor activity of the immune system. Iwafuchi et al. demonstrated that elevated PD-1/PD-L1 expression was associated with a poor prognosis in pediatric ALK+ ALCL 22. Three different case reports have described dramatic responses (CR, CR, CR) to PD-1 inhibitors in heavily pre-treated patients with R/R ALK+ ALCL. The combination of BV and NIVO has been extensively tested in both pediatric and adult patients with R/R Hodgkin lymphoma and R/R primary mediastinal B-cell lymphoma with robust safety and efficacy. Given the frequent expression of both CD30 and PD-L1 in ALK+ ALCL, the impressive single agent therapeutic efficacy of both BV and NIVO, and the tolerability of the combination of BV and NIVO in other patients with lymphoma, investigating the safety and efficacy of BV and NIVO in R/R ALK+ ALCL is warranted. For pediatric patients with relapsed or refractory ALK-positive ALCL, remission can be achieved through the use of chemotherapy and/or immune therapy. However, the optimal treatment strategy for consolidative therapy in pediatric patients with relapsed or refractory ALK- positive ALCL remains to be determined. The literature reports High-risk patients with CD3-positive ALCL experiencing relapse at any time after first-line therapy achieved 5-year EFS and OS rates of 62 and 73%, respectively after reinduction therapy followed by best available donor allogeneic stem cell transplantation. Very high-risk patients with progression during first-line therapy achieved EFS and OS rates of 41 and 59%, respectively after reinduction therapy followed by best available donor allogeneic stem cell transplantation. For all evaluable patients, the 5-year EFS and OS rates were 53 and 78%, respectively. A major barrier to survival for pediatric patients with relapsed or refractory ALCL is progression of disease during reinduction therapy prior to stem cell transplantation, highlighting the importance of effective re-induction therapy. Limited toxicity associated with immune therapy in comparison to traditional cytotoxic chemotherapy may contribute to more rapid recovery, reduction in time to stem cell transplantation and improvement in performance score prior to stem cell transplantation. Through the use of allogeneic stem cell transplantation and donor lymphocyte infusion, a graft versus lymphoma effect has been suggested for pediatric patients with relapsed or refractory ALCL.

ELIGIBILITY:
Inclusion Criteria:

* Patients must weigh ≥10 kilograms at the time of study enrollment.
* Patients with relapsed or refractory histologically or cytologically proven ALK-positive anaplastic large cell lymphoma.
* Patients must have adequate organ function.
* Patients must have performance status 60 or above.

Exclusion Criteria:

* ALK-NEGATIVE anaplastic large cell lymphoma.
* Patients with active leptomeningeal disease (lymphoma cells in CSF).
* Previous treatment with vinblastine (only in patients in the LR cohort).
* Female patients who are pregnant. Pregnancy tests must be obtained in girls who are post menarche.
* Lactating females unless they have agreed not to breastfeed their infants.
* Patients with Down syndrome.
* Any patient with uncontrolled infection prior to study entry.
* Any patient known to have primary or acquired immunodeficiency and/or prior solid organ transplant.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of adverse events (safety) of NIVO and Vinblastine (VBL) in CAYA with high-risk R/R ALK+ ALCL with prior exposure to Brentuximab vedotin (BV) | 1 year
  adverse events possible probably or definitely related to NIVO will be reported.
To determine the overall response rate of NIVO and Vinblastine (VBL) in CAYA with high-risk R/R ALK+ ALCL with prior exposure to Brentuximab vedotin (BV). | 1 year
  Patient will have disease assessments to determine best response to therapy with NIVO and Vinblastine
To determine the safety of NIVO and BV in CAYA with high-risk R/R ALK+ ALCL who have never received BV. | 1 year
  adverse events probably or definitely related to NIVO will be collected.
To determine the overall response rate to NIVO and BV in CAYA with high-risk R/R ALK+ ALCL who have never received BV. | 1 year
  disease assessments will be performed to determine best response post therapy
To significantly improve the 1 year EFS in CAYA with high-risk ALCL who received NIVO risk-adapted combining immunotherapy with re-induction followed by RTC and AlloHSCT compared to historical controls. | 1 year
  Events for EFS the first year will be reported and are defined as disease relapse, disease progression or toxic death.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No